CLINICAL TRIAL: NCT02776904
Title: Comprehensive Dynamic Movement Assessment for Concussion Management
Brief Title: Movement Assessment for Concussion Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 205006
Record Dates: First submitted 2016-05-17; First posted 2016-05-18 (Estimated); Results first posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Healthy Athlete
Keywords: Concussion; Football player; Movement assessment; Soccer player
MeSH Terms: conditions — Brain Concussion | interventions — Neuropsychological Tests; Gait; Single Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy athlete (Other): Healthy athletes (14-18 years old) enrolled in sports program in local schools.
  Interventions: Other: Immediate Post-concussion Assessment and Cognitive Testing; Other: Gait with single and dual task; Other: Y-Balance test; Other: Psychomotor Vigilance Task
- Concussed athletes (Other): Concussed athletes from a sports related injury who are 14-18 years old and referred to a regional sports concussion clinic.
  Interventions: Other: Gait with single and dual task; Other: Y-Balance test

INTERVENTIONS:
Other: Immediate Post-concussion Assessment and Cognitive Testing — Computerized assessment that provides information related to visual reaction time and visual memory.
  Other Names: ImPACT
  Arms: Healthy athlete
Other: Gait with single and dual task — Walking alone and then walking while performing a memory task on a tablet.
Other: Y-Balance test — Dynamic balance test measuring reaching of the leg to the anterior,postero- lateral, and postero-medial directions.
  Other Names: Star Excursion Balance Test (SEBT)
Other: Psychomotor Vigilance Task — Assessment measuring reaction time based on auditory cues.
  Other Names: PVT
  Arms: Healthy athlete

SUMMARY:
Previous work in the area of concussion management has focused heavily on neuro-cognitive testing. In addition to routine neuro-cognitive testing through Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT),this pilot study is designed to establish a comprehensive battery of clinical assessment through the utilization of functional movement and dynamic postural control assessments. The immediate application of these assessments will be focused on the male high school football player (who is at risk for concussion) and both female and male soccer players. Our pilot study aims determine the stability of ImPACT testing in youth athletes in light of ongoing neurodevelopment in this population. In addition, this pilot work will implement additional tools focused on assessment of dynamic balance and gait. This approach will significantly enhance predictions of subsequent musculoskeletal injuries that have been shown to occur in concussed collegiate and professional athletes and that we believe are also occurring in our high school athletes. This battery of tests will provide clinicians with invaluable information to guide both rehabilitation of and return to play (RTP) decisions for concussed high school athletes.

DETAILED DESCRIPTION:
Experiment 1. High school athletes will complete a battery of tests including the Y-balance test, a version of the Star Excursion Balance Test (SEBT), a divided attention gait task, the Psychomotor Vigilance Task (PVT). The SEBT is an established, reliable outcome measure of dynamic postural stability through measurement of lower extremity reach distance. Our study will also utilize a force plate during SEBT testing to allow the investigators to sensitively measure center of mass in all planes. To test gait balance control and adaptation of gait strategy which have been shown to be impaired in concussed individuals acutely and chronically, athletes will walk at self-selected speed on the GAITRite® portable gait analysis walkway for three undivided attention trials and three divided attention trials during which a cognitive task, will be imposed.The GaitRite® will calculate spatio-temporal parameters during gait and has been used in the concussion literature. The PVT is a reliable and valid measurement of simple reaction time to an auditory cue. The outcome measure will be the mean reaction time. These tests were administered by licensed physical therapists, assisted by students from both the Doctorate of Physical Therapy (DPT) and PhD physical therapy programs at UCA, before the initiation of summer 2016 football practices for all athletes in the program. The total testing time per athlete will not exceed 1.5 hours. The battery will be administered again to all athletes in the football program after the season has ended and prior to the end of the school year in the spring 2017. The 2017-2019 season will test both football and soccer (male and female athletes) and will include functional testing for athletes who have had a concussion through concussion clinic.

Experiment 2. Qualified athletic trainers or Physical Therapists, with oversight by Dr. Israel, will administer the ImPACT using the same schedule as described in Experiment 1. The ImPACT is a widely used neurocognitive testing component of the standard three-prong approach to concussion management which also includes symptom inventories and static balance assessment. The computerized test evaluates concentration, attention, memory, visual motor speed, and reaction time. High sensitivity and specificity for concussion using the ImPACT has been shown. The test also has been shown to be a valid and reliable measure in the high school and collegiate populations. Composite scores for each of the non-injured athletes will be stratified by age to examine changes across the three assessments. Hunt and Ferrara have shown significant change in baseline assessments between 9th grade and 11th and 12th grade age groups driven by 9th grade test scores indicating that biennial testing for young adolescents may not be sufficient.The current recommendation for this younger age group is annual testing, though recent studies call for the investigation of even more frequent testing, thus our plan to test at six months. ImPACT testing will not exceed 1 hour. The 2017-2018 season will test both football and soccer (male and female athletes) for ImPACT testing.

ELIGIBILITY:
Inclusion Criteria:

* Male football players (2016 and 2017 season)
* Male and female soccer players (2017-2018 and 2018-2019 season) OR Athletes who have been diagnosed with a sports related concussion during the season of their assigned sport and is being seen through concussion clinic at Arkansas children's hospital

  * Age 14-18
  * Written informed consent from the parent

Exclusion Criteria:

* Athletes who have not completed pre-participation physicals
* Any condition that the investigator determines would put the subject at risk if participating in the study.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Male football players and both male and female soccer players
Enrollment: 327 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Joe T. Robinson High School, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langlois JA, Rutland-Brown W, Wald MM. The epidemiology and impact of traumatic brain injury: a brief overview. J Head Trauma Rehabil. 2006 Sep-Oct;21(5):375-8. doi: 10.1097/00001199-200609000-00001. PMID 16983222

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Athletes: Healthy Adolescent school athletes 14-18 years old were recruited from central Arkansas schools to complete assessments of gait, balance and computerized cognitive testing through the ImPACT(Immediate post concussion assessment and cognitive testing) baseline assessment.
- Concussed Athletes: Adolescent males and females (14-19 years of age) with concussion who visited the concussion clinic at a regional Children's Hospital.
Period: Overall Study
Arm/Group | Healthy Athletes | Concussed Athletes
Started | 281 | 46
Gait Assessment | 178 | 32
ImPACT | 21 | 46 (ImPACT testing for the concussed subjects was completed for the clinical assessment (not research).)
Completed | 281 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Athletes | Concussed Athletes | Total
Number analyzed (Participants) | 281 | 46 | 327
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 281 | 46 | 327
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 17 | 133
  Male | 165 | 29 | 194
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 132 | 44 | 176
  African American | 108 | 1 | 109
  Two or More Races | 0 | 1 | 1
  Not Selected | 41 | 0 | 41

OUTCOME MEASURES:

1. Primary Outcome: Impact ( Immediate Post-concussion Assessment and Cognitive Testing) Healthy Athlete
Description: Verbal memory (total % correct from design memory, total correct from memory score from X's and O's) and visual memory (total number correct/4 during module 3) Scores on verbal memory and visual memory range from 70-99 (high scores are better than low scores).
  Visual motor speed is comprised correct responses/4 for specific modules and the average counted correctly x3 for a specific module.
  Scores range from 27-39.8 (high scores are better than low scores)
Time Frame: preseason, postseason, end of the school year, pre-season year 2
Population: subset from healthy athlete group
Measure: Mean (Standard Error); unit: score on Immediate post concussion scale
Groups:
- Healthy Athlete IMPACT Score: Immediate Post-concussion Assessment and Cognitive Testing will be administered three times (pre-season, post season and end of year) during the school year and testing will not exceed 1 hour per athlete.
  Immediate Post-concussion Assessment and Cognitive Testing
Arm/Group | Healthy Athlete IMPACT Score
Number analyzed (Participants) | 21
score on Immediate post concussion scale
  pre season verbal memory | 86.33 (1.470)
  post season year verbal memory | 84.0 (2.379)
  end of school verbal memory | 90.73 (2.095)
  pre-season year 2 verbal memory | 89.1436 (2.707)
  pre-season visual memory | 69.8361 (3.54)
  post season visual memory | 81.2 (2.5824)
  end of the school year visual memory | 81.4659 (2.98)
  pre-season year 2 visual memory | 82.2006 (2.26)
  preseason visual motor composite | 36.371 (2.007)
  post season visual motor | 36.727 (2.05)
  end of school visual motor | 38.897 (2.215)
  pre-season year 2 visual motor | 39.3035 (1.665)
Statistical Analysis 1: Comparison: Healthy Athlete IMPACT Score; Repeated measures ANOVA compared pre-season scores to post-season, end of the school year and pre-season year 2 for Visual Memory; Test type: Other; p = 0.0003, ANOVA — Adjustment with Tukey-Kramer; 3 DF
Statistical Analysis 2: Comparison: Healthy Athlete IMPACT Score; Repeated measures ANOVA compared pre-season scores to post-season, end of the school year and pre-season year 2 for Verbal memory; Test type: Other; p = 0.0281, ANOVA — Adjusted for multiple comparisons using Tukey-Kramer; DF 3
Statistical Analysis 3: Comparison: Healthy Athlete IMPACT Score; Repeated measures ANOVA compared pre-season scores to post-season, end of the school year and pre-season year 2 for Visual Motor composite; Test type: Other; p = 0.0035, ANOVA — Adjusted for multiple comparisons; DF 3

2. Primary Outcome: Impact ( Immediate Post-concussion Assessment and Cognitive Testing) Healthy Athlete
Description: Reaction time Composite is the average correct reaction time of 3 skills Scores range from 0.5 to 0.7 Lower scores are better.
Time Frame: preseason, postseason and end of the school year and preseason the following year
Population: subset from healthy athlete group Measured on Reaction time composite score (Immediate Post Concussion Assessment)
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Healthy Athlete IMPACT Score
Number analyzed (Participants) | 21
seconds
  Preseason | 0.5797 (0.016)
  Post Season | 0.5780 (0.01615)
  End of the school year | 0.5902 (0.0166)
  Pre-season year 2 | 0.6089 (0.01792)
Statistical Analysis 1: Comparison: Healthy Athlete IMPACT Score; Repeated measures ANOVA compared pre-season scores to post-season, end of the school year and pre-season year 2 for Reaction Time; Test type: Other; p = 0.2637, ANOVA — Adjusted for multiple comparisons using Tukey-Kramer

3. Primary Outcome: Spatiotemporal Gait Parameters- Gait Velocity
Description: For the purposes of this study, parameters that were captured by the GAITRite® include: gait velocity (cm/s); Subjects walk on pathway during single task and dual task is walking while performing a visual memory task on a tablet
Time Frame: Cross-sectional baseline
Population: Data are not mutually exclusive. Reported for single task and dual task and divided into male and female groups.
Measure: Mean (Standard Deviation); unit: cm/sec
Groups:
- Gait Assessment- Velocity: Gait parameters were assessed by instructing the participants to walk at a self-selected speed on the GAITRite® (CIR Systems, Inc.; Franklin, NJ) portable gait analysis walkway for three, undivided attention trials and three, divided attention trials. During each divided attention trial, a visuospatial memory task was given to the subjects to complete on a tablet (Microsoft Surface Pro, 2016) while walking. The GAITRite® portable gait analysis walkway and corresponding GAITRite® software recorded temporal and spatial parameters. Prior to each participant's trials, investigators entered leg length data. Leg length was measured as the distance from greater trochanter to floor for each leg. For the purposes of this study, parameters that were captured by the GAITRite® include: gait velocity (cm/s); step length (cm); DLS, defined as the percent of the gait cycle (%GC) when both feet are on the ground; and SLS, defined as the %GC weight bearing through a single limb.
Arm/Group | Gait Assessment- Velocity
Number analyzed (Participants) | 210
cm/sec
  Single Task Gait Velocity Male: number analyzed (Participants) | 128
  Single Task Gait Velocity Male | 1.236 (0.163)
  Single Task Gait Velocity Female: number analyzed (Participants) | 50
  Single Task Gait Velocity Female | 1.449 (0.199)
  Dual Task Gait Velocity Male: number analyzed (Participants) | 128
  Dual Task Gait Velocity Male | 1.030 (0.185)
  Dual Task Gait Velocity Female: number analyzed (Participants) | 50
  Dual Task Gait Velocity Female | 1.232 (0.196)
  Single Task Gait Velocity Female Concussed: number analyzed (Participants) | 14
  Single Task Gait Velocity Female Concussed | 1.207 (0.238)
  Dual Task Gait Velocity Female Concussed: number analyzed (Participants) | 14
  Dual Task Gait Velocity Female Concussed | 0.974 (0.18)
  Single Task Gait Velocity Male Concussed: number analyzed (Participants) | 18
  Single Task Gait Velocity Male Concussed | 1.125 (0.14)
  Dual Task Gait Velocity Male Concussed: number analyzed (Participants) | 18
  Dual Task Gait Velocity Male Concussed | 0.922 (0.18)
Statistical Analysis 1: Comparison: Gait Assessment- Velocity; Descriptive analysis, including means and standard deviations was used to summarize all participant data. Velocity was normalized to leg length. Normality was tested and assumed for all measured gait parameters for healthy athletes. A two-way repeated measure analyses of variance (ANOVA) was used to explore the impact of walk status and sex on gait velocity for healthy athletes. Adjusted using Tukey's post hoc method for the pairwise comparisons (0.05 threshold for significance); Test type: Other; p < 0.001, ANOVA — Used Tukey's Adjustment

4. Primary Outcome: Gait Parameters: Step Length (Cm)
Description: For the purposes of this study, parameters that were captured by the GAITRite® include:step length (cm);
Time Frame: cross-sectional baseline
Population: Data are not mutually exclusive. Reported for single task and dual task and divided into male and female groups and healthy and concussed athletes
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Gait Assessment: Gait parameters were assessed by instructing the participants to walk at a self-selected speed on the GAITRite® (CIR Systems, Inc.; Franklin, NJ) portable gait analysis walkway for three, undivided attention trials and three, divided attention trials. During each divided attention trial, a visuospatial memory task was given to the subjects to complete on a tablet (Microsoft Surface Pro, 2016) while walking. The GAITRite® portable gait analysis walkway and corresponding GAITRite® software recorded temporal and spatial parameters. Prior to each participant's trials, investigators entered leg length data. Leg length was measured as the distance from greater trochanter to floor for each leg. For the purposes of this study, parameters that were captured by the GAITRite® include: step length (cm)
Arm/Group | Gait Assessment
Number analyzed (Participants) | 210
cm
  Single task step length males: number analyzed (Participants) | 128
  Single task step length males | 68.031 (6.779)
  Single task step length female: number analyzed (Participants) | 50
  Single task step length female | 65.483 (6.021)
  Dual Task Step Length Male: number analyzed (Participants) | 128
  Dual Task Step Length Male | 60.073 (7.858)
  Dual Task Step Length Female: number analyzed (Participants) | 50
  Dual Task Step Length Female | 58.650 (5.885)
  Single Task Step Length Female concussed: number analyzed (Participants) | 14
  Single Task Step Length Female concussed | 61.26 (7.94)
  Dual Task Gait step length Female Concussed: number analyzed (Participants) | 14
  Dual Task Gait step length Female Concussed | 57.22 (12.79)
  Single Task Step length Male Concussed: number analyzed (Participants) | 18
  Single Task Step length Male Concussed | 65.63 (5.11)
  Dual Task Step length Male Concussed: number analyzed (Participants) | 18
  Dual Task Step length Male Concussed | 57.71 (6.37)
Statistical Analysis 1: Comparison: Gait Assessment; Test type: Other — Normality was tested and assumed for all measured gait parameters. A two-way repeated measure analyses of variance (ANOVA) was used to explore the impact of walk status and sex on gait parameters of step length. Adjusted using Tukey's post hoc method for the pairwise comparisons (0.05 threshold for significance); p < 0.0001, ANOVA; Tukey's post hoc method for the pair wise comparisons between walk status and sex for step length

5. Primary Outcome: Gait Parameters- Percent of DLS
Description: DLS, defined as the percent of the gait cycle (%GC) when both feet are on the ground measured in healthy males and female athletes and concussed males and female athletes
Time Frame: cross-sectional baseline
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of GC spent on 2 limbs
Groups:
- Gait Assessment- DLS: Gait parameters were assessed by instructing the participants to walk at a self-selected speed on the GAITRite® (CIR Systems, Inc.; Franklin, NJ) portable gait analysis walkway for three, undivided attention trials and three, divided attention trials. During each divided attention trial, a visuospatial memory task was given to the subjects to complete on a tablet (Microsoft Surface Pro, 2016) while walking. The GAITRite® portable gait analysis walkway and corresponding GAITRite® software recorded temporal and spatial parameters. Prior to each participant's trials, investigators entered leg length data. Leg length was measured as the distance from greater trochanter to floor for each leg. For the purposes of this study, parameters that were captured by the GAITRite® include: gait velocity (cm/s); step length (cm); DLS, defined as the percent of the gait cycle (%GC) when both feet are on the ground; and SLS, defined as the %GC weight bearing through a single limb.
Arm/Group | Gait Assessment- DLS
Number analyzed (Participants) | 210
percentage of GC spent on 2 limbs
  Single task % GC in DLS Male: number analyzed (Participants) | 128
  Single task % GC in DLS Male | 29.077 (2.631)
  Single task % GC in DLS Female: number analyzed (Participants) | 50
  Single task % GC in DLS Female | 26.922 (2.648)
  Dual task % GC in DLS Male: number analyzed (Participants) | 128
  Dual task % GC in DLS Male | 31.92 (3.461)
  Dual task % GC in DLS Females: number analyzed (Participants) | 50
  Dual task % GC in DLS Females | 29.542 (3.085)
  Single Task % GC in DLS Female Concussed: number analyzed (Participants) | 14
  Single Task % GC in DLS Female Concussed | 28.09 (3.66)
  Dual Task % of GC in DLS Female: number analyzed (Participants) | 14
  Dual Task % of GC in DLS Female | 30.45 (5.29)
  Single task % of GC in DLS male concussed: number analyzed (Participants) | 18
  Single task % of GC in DLS male concussed | 30.33 (2.13)
  Dual Task % GC in DLS Male Concussed: number analyzed (Participants) | 18
  Dual Task % GC in DLS Male Concussed | 32.32 (2.66)
Statistical Analysis 1: Comparison: Gait Assessment- DLS; Test type: Other — Normality was tested and assumed for all measured gait parameters. A two-way repeated measure analyses of variance (ANOVA) was used to explore the impact of walk status and sex on percent of gait cycle in DLS; p < 0.0001, ANOVA; Tukey's post hoc method for the pairwise comparisons with p<.05

6. Primary Outcome: Gait Parameters- % of Gait Cycle in SLS
Description: For the purposes of this study, parameters that were captured by the GAITRite® include: SLS, defined as the %GC weight bearing through a single limb.
Time Frame: cross-sectional baseline
Population: Data are not mutually exclusive. Reported for single task and dual task and divided into male and female groups as well as healthy and concussed athletes.
Measure: Mean (Standard Deviation); unit: percentage of gait cycle spent on 1 limb
Groups:
- Gait Assessment- SLS Healthy Athlete: Gait parameters were assessed by instructing the participants to walk at a self-selected speed on the GAITRite® (CIR Systems, Inc.; Franklin, NJ) portable gait analysis walkway for three, undivided attention trials and three, divided attention trials. During each divided attention trial, a visuospatial memory task was given to the subjects to complete on a tablet (Microsoft Surface Pro, 2016) while walking. The GAITRite® portable gait analysis walkway and corresponding GAITRite® software recorded temporal and spatial parameters. Prior to each participant's trials, investigators entered leg length data. Leg length was measured as the distance from greater trochanter to floor for each leg. For the purposes of this study, parameters that were captured by the GAITRite® include: SLS, defined as the %GC weight bearing through a single limb.
Arm/Group | Gait Assessment- SLS Healthy Athlete
Number analyzed (Participants) | 210
percentage of gait cycle spent on 1 limb
  Single task % GC in SLS Male: number analyzed (Participants) | 128
  Single task % GC in SLS Male | 35.290 (1.504)
  Single task % GC in SLS Female: number analyzed (Participants) | 50
  Single task % GC in SLS Female | 36.522 (1.352)
  Dual task % GC in SLS Male: number analyzed (Participants) | 128
  Dual task % GC in SLS Male | 34.05 (1.901)
  Dual task % GC in SLS Females: number analyzed (Participants) | 50
  Dual task % GC in SLS Females | 35.112 (1.549)
  Single Task % GC Female Concussed: number analyzed (Participants) | 14
  Single Task % GC Female Concussed | 35.85 (1.796)
  Dual Task % GC Female Concussed: number analyzed (Participants) | 14
  Dual Task % GC Female Concussed | 34.407 (1.974)
  Single task % of GC in SLS male concussed: number analyzed (Participants) | 18
  Single task % of GC in SLS male concussed | 34.62 (1.03)
  Dual Task % GC in SLS Male Concussed: number analyzed (Participants) | 18
  Dual Task % GC in SLS Male Concussed | 33.58 (1.26)
Statistical Analysis 1: Comparison: Gait Assessment- SLS Healthy Athlete; Test type: Other — Normality was tested and assumed for all measured gait parameters. A two-way repeated measure analyses of variance (ANOVA) was used to explore the impact of walk status and sex on percent of gait cycle in SLS; p < 0.0001, ANOVA; Tukey's post hoc method for pairwise comparison between walk status and sex for %GC in SLS

7. Primary Outcome: Y Balance Assessment- Anterior Reach Direction
Description: subset from healthy athlete group and concussed group Measured on YBT in anterior direction
Time Frame: Cross sectional baseline
Population: Data are not mutually exclusive. Reported for Y balance test divided into male and female groups. Data for concussed subjects is reported in the acute phase and divided into male and female groups.
Measure: Mean (Standard Deviation); unit: Index
Groups:
- Y Balance Data: Y balance data anterior reach distance (cm) normalized to leg length (cm) [(reach distance/leg length) x 100] providing an index value of the normalized reach distance.
Arm/Group | Y Balance Data
Number analyzed (Participants) | 212
Index
  Male healthy athletes: number analyzed (Participants) | 111
  Male healthy athletes | 95.34 (10.814)
  Female healthy athletes: number analyzed (Participants) | 69
  Female healthy athletes | 94.45 (14.52)
  male acute concussed: number analyzed (Participants) | 22
  male acute concussed | 95.13 (9.8)
  female acute concussed: number analyzed (Participants) | 10
  female acute concussed | 95.14 (12.48)
Statistical Analysis 1: Comparison: Y Balance Data; Test type: Other; p > 0.05, ANOVA

8. Primary Outcome: Y Balance Assessment- Posterolateral Reach Direction
Description: subset from healthy athlete group and concussed group Measured on YBT in postero-lateral direction.
Time Frame: Cross sectional baseline
Population: Data are not mutually exclusive. Reported for Y balance test divided into male and female groups and healthy and concussed athletes. Data for concussed subjects is reported in the acute phase and divided into male and female groups.
Measure: Mean (Standard Deviation); unit: Index
Groups:
- Y Balance Data: Y balance data posterolateral reach distance (cm) normalized to leg length (cm) [(reach distance/leg length) x 100] providing an index value of the normalized reach distance in the posterolateral direction.
Arm/Group | Y Balance Data
Number analyzed (Participants) | 212
Index
  Male healthy athletes: number analyzed (Participants) | 111
  Male healthy athletes | 78.08 (10.697)
  Female healthy athletes: number analyzed (Participants) | 69
  Female healthy athletes | 70.138 (10.120)
  Male acute concussed: number analyzed (Participants) | 22
  Male acute concussed | 74.21 (10.44)
  female acute concussed: number analyzed (Participants) | 10
  female acute concussed | 83.89 (14.14)
Statistical Analysis 1: Comparison: Y Balance Data; Test type: Other; p > 0.05, ANOVA

9. Primary Outcome: Y Balance Assessment- Postero-medial Reach Direction
Description: subset from healthy athlete group and concussed group Measured on YBT in postero-medial direction.
Time Frame: Cross sectional baseline
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Index
Groups:
- Y Balance Data: Y balance data postero-medial reach distance (cm) normalized to leg length (cm) [(reach distance/leg length) x 100] providing an index value of the normalized reach distance.
Arm/Group | Y Balance Data
Number analyzed (Participants) | 212
Index
  Male healthy athletes: number analyzed (Participants) | 111
  Male healthy athletes | 69.750 (12.590)
  Female healthy athletes: number analyzed (Participants) | 69
  Female healthy athletes | 65.860 (8.768)
  male acute concussed: number analyzed (Participants) | 22
  male acute concussed | 68.80 (11.13)
  female acute concussed: number analyzed (Participants) | 10
  female acute concussed | 69.17 (12.66)
Statistical Analysis 1: Comparison: Y Balance Data; Test type: Other; p > 0.05, ANOVA

10. Primary Outcome: Psychomotor Vigilance Task (PVT)
Description: The PVT is a reliable and valid measurement of simple reaction time to an auditory cue. The outcome measure will be the mean reaction time.
Time Frame: cross-sectional baseline
Population: Subset of healthy athletes. The Concussed athlete data for the PVT (as was the ImPACT concussed data) was used clinically to assess individual auditory reaction time and for clinical decision making by the medical team. The concussed PVT data will not be used as aggregate data.
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Healthy Athlete PVT Score: PVT testing will occur during a session of baseline testing in healthy male athletes who are participating in high school sports.
Arm/Group | Healthy Athlete PVT Score
Number analyzed (Participants) | 105
ms | 218.57 (62.78)

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- Healthy Athletes: Healthy athletes were assessed using Gait analysis, balance, and ImPACT in their schools.
- Concussed Athletes: concussed athletes were assessed using Gait Analysis, balance, and IMPACT.
Arm/Group | Healthy Athletes | Concussed Athletes
All-Cause Mortality (participants affected / at risk) | 0/281 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/281 | 0/46
Other Adverse Events (participants affected / at risk) | 0/281 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT02776904/Prot_SAP_000.pdf